CLINICAL TRIAL: NCT04945460
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of Sotatercept Versus Placebo for the Treatment of Combined Postcapillary and Precapillary Pulmonary Hypertension (Cpc-PH) Due to Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: A Study of Sotatercept for the Treatment of Cpc-PH Due to HFpEF (MK-7962-007/A011-16)
Acronym: CADENCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7962-007; A011-16 (Other: Acceleronpharma); MK-7962-007 (Other: MSD); 2023-509141-12-00 (Registry Identifier: EU CT); U1111-1309-6433 (Registry Identifier: UTN); 2021-003020-32 (EudraCT Number)
Record Dates: First submitted 2021-06-11; First posted 2021-06-30 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary, hypertension, Cpc PH, HFpEF, sotatercept
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension | interventions — ACE-011

STUDY DESIGN:
Intervention Model Description: Each eligible participant will be randomly assigned in a 1:1:1 ratio to 1 of the 3 treatment groups during the Treatment Period:
  Arm 1: Treatment Group 1: Placebo delivered subcutaneously (SC) every 3 weeks (Q3W) for 24 weeks
  Arm 2: Treatment Group 2: Sotatercept SC at a dose level of 0.3 mg/kg Q3W for 24 weeks
  Arm 3: Treatment Group 3: Sotatercept SC at a starting dose level of 0.3 mg/kg for 3 dosing visits (Q3W), then escalating to 0.7 mg/kg SC on the fourth dosing visit and Q3W for the remainder of the 24-week Treatment Period
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Delivered subcutaneously (SC) every 3 weeks (Q3W) for 24 weeks in the placebo-controlled treatment period.
  Interventions: Drug: Placebo
- Sotatercept 0.3 mg/kg (Experimental): Participants will receive sotatercept SC at a dose level of 0.3 mg/kg Q3W for 24 weeks in the placebo-controlled treatment period.
  Interventions: Drug: Sotatercept 0.3 mg/kg
- Sotatercept 0.3 mg/kg, escalating to 0.7 mg.kg (Experimental): Sotatercept SC at a starting dose level of 0.3 mg/kg for 3 dosing visits (Q3W), then escalating to 0.7 mg/kg SC on the fourth dosing visit and Q3W for the remainder of the 24-week treatment Period.
  Interventions: Drug: Sotatercept 0.3 mg/kg escalating to 0.7 mg/kg

INTERVENTIONS:
Drug: Sotatercept 0.3 mg/kg — Administered by subcutaneous injection. Sotatercept (ACE-011) is a recombinant fusion protein consisting of the extracellular domain of the human activin receptor type IIA linked to the Fc piece of human IgG1.
  Other Names: ACE-011
  Arms: Sotatercept 0.3 mg/kg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo
Drug: Sotatercept 0.3 mg/kg escalating to 0.7 mg/kg — Administered by subcutaneous injection. Sotatercept (ACE-011) is a recombinant fusion protein consisting of the extracellular domain of the human activin receptor type IIA linked to the Fc piece of human IgG1.
  Other Names: ACE-011
  Arms: Sotatercept 0.3 mg/kg, escalating to 0.7 mg.kg

SUMMARY:
This is a Phase 2, double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of sotatercept versus placebo in adults with Cpc-PH due to HFpEF.

The objective of this study is to evaluate the efficacy, safety and tolerability of sotatercept versus placebo in adults with Cpc-PH due to HFpEF. Efficacy is measured by change from baseline in pulmonary vascular resistance (PVR, primary endpoint) and 6-minute walk distance (6MWD, key secondary endpoint).

DETAILED DESCRIPTION:
Participants enrolled in the study will have a diagnosis of Cpc-PH due to HFpEF with New York Heart Association (NYHA) functional class (FC) II or III. Participants will be randomly assigned in a 1:1:1 ratio to 1 of the 3 treatment groups (placebo, 0.3mg/kg sotatercept and 0.7mg/kg sotatercept) during the placebo-controlled Treatment Period. In the extension phase, sotatercept-treated participants will continue on their current dose. Placebo participants will be re-randomized in a 1:1 ratio to one of the two sotatercept treatment groups utilized in the placebo-controlled Treatment Period. Each participant will be enrolled in the study for up to 114 weeks, including a 28-day Screening Period, a 24-week, double-blind, placebo-controlled Treatment Period, an 18-month Extension Period, and an 8-week Follow-up Period.

As of protocol amendment 6, the 18-month Extension Period is being removed. Participants who have completed at least the 24-week placebo controlled treatment period and the end of study visit, and who have not discontinued study treatment early, may be eligible to participate in an extension study.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be enrolled in this proof-of-concept study:

1. Age 18 to 85 years
2. Clinical diagnosis of HFpEF:

   • Left ventricular ejection fraction ≥50%, with no history of LVEF below 45% in more than two consecutive measurements under stable conditions
3. Demonstrated Cpc-PH by all of the following:

   * Baseline RHC performed within 28 days of randomization documenting a minimum PVR of ≥320 dyn•sec/cm5 (4 wood units)
   * Mean pulmonary arterial pressure (mPAP) of >20 mmHg
   * Pulmonary capillary wedge pressure (PCWP) >15 mmHg but < 30 mmHg
4. New York Heart Association FC of II or III
5. Six-minute Walk Distance ≥100 m repeated twice during Screening and both values within 15% of each other, calculated from the highest value
6. Chronic medication for HF or for any underlying condition, administered at a stable (per investigator) dose for ≥30 days prior to Visit 1. Diuretics and/or anticoagulants are excepted from this rule but should not be newly started or stopped within 30 days of Visit 1, and a prescribed dose change should not occur within 7 days of Visit 1. Anticoagulation may be suspended for RHC if necessary.
7. Women of childbearing potential must:

   * Have 2 negative urine or serum pregnancy tests as verified by the investigator during the Screening Period; must agree to ongoing pregnancy testing during the course of the study and until 8 weeks after the last dose of the study drug
   * If sexually active with a male partner: use highly effective contraception without interruption for at least 28 days prior to starting the investigational product AND agree to use the same highly effective contraception in combination with a barrier method during the study (including dose interruptions), and for 16 weeks (112 days) after discontinuation of study treatment
   * Refrain from breastfeeding a child or donating blood, eggs, or ovum for the duration of the study and for at least 16 weeks (112 days) after the last dose of study drug
8. Male participants must:

   * Agree to use a condom, defined as a male latex condom or non latex condom NOT made out of natural (animal) membrane (e.g., polyurethane), during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for at least 16 weeks (112 days) following investigational product discontinuation, even if he has undergone a successful vasectomy
   * Refrain from donating blood or sperm for the duration of the study and for 16 weeks (112 days) after the last dose of study drug
9. Ability to adhere to the study visit schedule and understand and comply with all protocol requirements
10. Agreement to not participate in any other trials of investigational drugs/devices while enrolled in the A011-16 study
11. Ability to understand and provide documented consent for participation

Exclusion Criteria:

Participants will be excluded from the study if any of the following criteria are met:

1. A diagnosis of PH in WHO Group 1, WHO Group 3, WHO Group 4, or WHO Group 5
2. Clinically significant and active lung disease:

   * Chronic obstructive pulmonary disease with post-bronchodilator forced expiratory volume in the first second (FEV1) <60% predicted
   * Restrictive lung disease with total lung capacity <70% predicted
   * More than mild interstitial lung disease (ILD), with FVC<70% or FEV1<60% predicted (still appropriate if absence of more than mild ILD, fibrosis, or COPD on computed tomography [CT] imaging)
3. Cardiovascular co-morbidities, which include any of the following:

   * History of more than mild mitral or aortic stenosis
   * Ongoing more than mild mitral or aortic regurgitation
   * More than one valve replacement or repair (mechanical or biomechanical) or anticipation of any valve replacement or repair
   * Severe tricuspid regurgitation due to primary valvular disease
   * Occurrence of myocardial infarction, acute coronary syndrome, coronary artery bypass graft or percutaneous coronary intervention within 180 days of Visit 1
   * History of serious life-threatening or hemodynamically significant arrhythmia
   * History of or anticipated heart transplant or ventricular assist device implantation
   * History of implantable cardioverter defibrillator placement or anticipated implantation of pacemaker, pacemaker implantation within 30 days of Screening
   * Anticipated implantation of pacemaker, pacemaker implantation within 30 days of Screening or history of implantable cardioverter defibrillator placement
   * Occurrence of myocardial infarction within 180 days of Visit 1
   * History of known pericardial constriction, hypertrophic cardiomyopathy, sarcoidosis, or amyloid cardiomyopathy
   * Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure >160 mmHg or sitting diastolic blood pressure >110 mmHg during Screening after a period of rest
   * Systemic hypotension as evidenced by sitting systolic blood pressure <90 mmHg or sitting diastolic blood pressure <50 mmHg during Screening
   * Resting heart rate of <45 bpm or >115 bpm
   * Stroke within 90 days of Visit 1
   * Acutely decompensated HF that required hospitalization within 30 days of Visit 1
   * Electrocardiogram during Screening Period with Fridericia's corrected QT interval (QTcF) >470 msec for males or >480 msec for females, or >500 msec if a ventricular conduction defect (right bundle branch block; left bundle branch block; or interventricular conduction delay) is present
   * Personal or family history of Brugada syndrome, sudden cardiac arrest or unexplained sudden cardiac death or arrest
   * Personal or family history of long QT syndrome unless the participant's ECG shows a normal QTc
   * Arrhythmogenic right ventricular dysplasia (ARVD) unless the participant has a recent cardiac MRI that shows no evidence of this diagnosis
4. Hospitalization for any worsening of medical conditions or any significant surgery per investigator within 30 days of Visit 1.
5. Received any approved PAH-specific therapies (i.e., endothelin receptor antagonists, prostacyclin analogs, phosphodiesterase-5 inhibitors, soluble guanylate cyclase stimulators) within 30 days of Visit 1.The use of an oral phosphodiesterase type 5 inhibitor, if only indicated for erectile dysfunction, is permitted, if not administered within 48 hours of a study visit or procedure.
6. Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin,or levosimendan) within 30 days of Visit 1
7. Received erythropoietin within 6 months of Visit 1.
8. Known history of chronic liver disease, including untreated hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), with severe hepatic impairment and/or cirrhosis (e.g., hepatic encephalopathy)
9. Prior exposure to sotatercept or luspatercept.
10. Currently enrolled in or have completed any other investigational product study within 30 days for small molecule drugs or within 5 half-lives for investigational biologics prior to the date of documented consent.
11. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days of Visit 1 or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible).
12. Any of the following clinical laboratory values prior to Visit 1 as specified:

    * Hemoglobin (Hgb) above the gender-specific upper limit of normal (ULN) per local laboratory test within 28 days of Visit 1or <10 g/dL per local laboratory within 28 days of Visit 1
    * Serum alanine aminotransferase or aspartate aminotransferase levels >3× ULN or total bilirubin >3× ULN within 28 days of Visit 1
    * Estimated glomerular filtration rate <30 ml/min/1.73 m2 (4-variable Modification of Diet in Renal Disease equation) within 28 days of Visit 1 or required renal replacement therapy within 90 days of Visit 1
    * Glycated hemoglobin (HbA1c) >10% within 28 days of Visit 1
    * Platelet count < 75,000/mm3 within 28 days of Visit 1
13. History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients in the investigational product .
14. Major surgery within 60 days of Visit 1. Participants must have completely recovered from any previous surgery prior to Visit 1.
15. Prior organ transplantation (e.g., heart, lung, liver, kidney), bone marrow transplantation, or life expectancy of < 12 months.
16. Pregnancy or breastfeeding in females.
17. Active malignancy, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in situ, or ≤ 2 squamous cell carcinomas of the skin.
18. History of clinically significant (as determined by the investigator) endocrine, hematologic, hepatic, (auto)immune, infectious (requiring chronic antibiotics), metabolic, urologic, pulmonary, neurologic, neuromuscular, dermatologic, psychiatric, renal, and/or another disease that may limit participation in the study.
19. Body mass index ≥50 kg/m2.
20. More than mild obstructive sleep apnea (treated or untreated).
21. Any non-cardiopulmonary condition or acute/chronic impairment(s) (other than dyspnea) that limits the ability to perform 6-minute walk test (6MWT).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week 24 | Baseline and Week 24
  PVR, a hemodynamic variable of pulmonary circulation, is measured by right heart catheterization (RHC).

SECONDARY OUTCOMES:
Change From Baseline in the 6-Minute Walk Distance (6MWD) at Week 24 | Baseline and Week 24
  The 6MWD tests the distance walked in 6 minutes as a measure of functional capacity.
Time to First Clinical Worsening Event (TTCW) at Weeks 24 | Week 24
  Clinical Worsening events are defined as the number of weeks from first dose date to any of the following:
  * Hospitalization due to a cardiopulmonary indication (a non-elective hospitalization lasting at least 24 hours in duration caused by clinical conditions directly related to Pulmonary Hypertension and/or Heart Failure)
  * Administration of intravenous diuretics or subcutaneous (SC) furosemide
  * Death (all causes)
  * Decrease in 6 minute walk distance (6MWD) by ≥ 15% from baseline confirmed by 2 tests at least 4 hours, but no more than 1 week apart.
Change From Baseline in Mean Pulmonary Arterial Pressure (mPAP) at Week 24 | Baseline and Week 24
  mPAP is calculated from systolic and diastolic pulmonary artery pressure measured by right heart catheterization.
Change From Baseline in Pulmonary Capillary Wedge Pressure (PCWP) at Week 24 | Baseline and Week 24
  PCWP is an indirect estimate of left atrial pressure measured in right heart catheterization.
Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE) at Week 24 | Baseline and Week 24
  TAPSE is an echocardiographic measurement of tricuspid valve annulus movement, as an indicator of right heart function.
Change From Baseline in Right Ventricular Fractional Area Change (RVFAC) at Week 24 | Baseline and Week 24
  RVFAC is an echocardiographic measurement of percent change between right ventricular area during diastole and systole, as an indicator of right heart function.
Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Week 24 | Baseline and Week 24
  LVEF is an echocardiographic measurement of percent change between left ventricular volume during diastole and systole, as an indicator of left heart function.
Change From Baseline in Isovolumic Relaxation Time (IVRT) at Week 24 | Baseline and Week 24
  IVRT is an echocardiographic measurement of the interval between closure of the aortic valve, to onset of filling by opening of the mitral valve. It is used as an indicator of diastolic dysfunction.
Change From Baseline in ratio of mitral inflow velocity I to mitral annular velocity'(e') (E/e' ratio) at Week 24 | Baseline and Week 24
  E/e' is a ratio measured in echocardiography as an indicator of diastolic function.
Change From Baseline in the Ratio of the Peak Velocity Flow of the E Wave in Early Diastole to Peak Velocity Flow of the A Wave in Late Diastole (E/A Ratio) at Week 24 | Baseline and Week 24
  E/A is a ratio measured in echocardiography as an indicator of diastolic function.
Change From Baseline in N-terminal Pro-hormone Brain Natriuretic Peptide (NT-proBNP) at Week 24 | Baseline and Week 24
  NT-proBNP is a circulating biomarker that reflects myocardial stretch.
Change From Baseline in New York Heart Association Functional Class (NYHA FC) at Week 24 | Baseline and Week 24
  NYHA FC classifies the extent of heart failure.
Change From Baseline in Myocardial Contraction Fraction (MCF) at Week 24 | Baseline and Week 24
  MCF is an echocardiographic measurement that determines the ratio of left ventricular stroke volume to myocardial volume and is an indicator of left ventricular systolic function.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (119):
- United States (56):
  - PULMONARY ASSOCIATES, P.A. ( Site 1008), Phoenix, Arizona
  - University of Arizona ( Site 1006), Tucson, Arizona
  - Scripps Clinic ( Site 4001), La Jolla, California
  - Cedars Sinai Medical Center ( Site 1082), Los Angeles, California
  - University of California Irvine ( Site 1086), Orange, California
  - Jeffrey S.Sager MD Medical Corporation ( Site 1060), Santa Barbara, California
  - Stanford University ( Site 1024), Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center ( Site 1028), Torrance, California
  - University Of Colorado ( Site 1013), Aurora, Colorado
  - South Denver Cardiology Associates ( Site 1091), Littleton, Colorado
  - Winchester Chest Clinic ( Site 1093), New Haven, Connecticut
  - The George Washington University Medical Faculty Associates ( Site 1025), Washington D.C., District of Columbia
  - Bay Area Cardiology ( Site 1071), Brandon, Florida
  - Mayo Clinic Jacksonville - PPDS ( Site 1045), Jacksonville, Florida
  - AdventHealth Orlando ( Site 1058), Orlando, Florida
  - Tampa General Hospital ( Site 1043), Tampa, Florida
  - Piedmont Atlanta Hospital ( Site 1085), Atlanta, Georgia
  - Emory University ( Site 1030), Atlanta, Georgia
  - Saint Alphonsus Regional Medical Center ( Site 1097), Boise, Idaho
  - University of Illinois Hospital ( Site 1095), Chicago, Illinois
  - IU Health Advanced Heart and Lung Care ( Site 1092), Indianapolis, Indiana
  - Ascension Medical Group St. Vincent ( Site 1076), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 1050), Iowa City, Iowa
  - University of Kansas Medical Center ( Site 1020), Kansas City, Kansas
  - Norton Pulmonary Specialists ( Site 1066), Louisville, Kentucky
  - University of Louisville ( Site 1099), Louisville, Kentucky
  - University Medical Center New Orleans ( Site 1057), New Orleans, Louisiana
  - Tufts Medical Center - PPDS ( Site 1012), Boston, Massachusetts
  - Brigham and Women's Hospital [Boston, MA] ( Site 1014), Boston, Massachusetts
  - University of Michigan ( Site 1011), Ann Arbor, Michigan
  - University of Minnesota Hospitals ( Site 1062), Minneapolis, Minnesota
  - Washington University School of Medicine [Saint Louis, MO] ( Site 1022), St Louis, Missouri
  - University of Nebraska Medical Center ( Site 1053), Omaha, Nebraska
  - Pulmonary Health Physicians ( Site 1080), Liverpool, New York
  - Weill Cornell Medical College ( Site 1046), New York, New York
  - University of Rochester Medical Center - PPDS ( Site 1039), Rochester, New York
  - Duke University Medical Center ( Site 1026), Durham, North Carolina
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital ( Site 1001), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 1005), Cleveland, Ohio
  - Cleveland Clinic Foundation ( Site 1065), Cleveland, Ohio
  - The Ohio State University Wexner Medical Center ( Site 1032), Columbus, Ohio
  - University of Toledo Medical Center ( Site 1070), Toledo, Ohio
  - Oregon Health Science University ( Site 1054), Portland, Oregon
  - Allegheny General Hospital ( Site 1088), Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research ( Site 1089), Wynnewood, Pennsylvania
  - Rhode Island Hospital ( Site 1033), Providence, Rhode Island
  - Medical University of South Carolina - PPDS ( Site 1003), Charleston, South Carolina
  - Statcare Pulmonary Consultants - Knoxville ( Site 1031), Knoxville, Tennessee
  - Baylor University Medical Center ( Site 1096), Dallas, Texas
  - University of Texas Southwestern Medical Center ( Site 4002), Dallas, Texas
  - Intermountain Medical Center ( Site 1079), Murray, Utah
  - Inova Heart and Vascular Institute ( Site 1078), Falls Church, Virginia
  - Bon Secours St. Mary's Hospital ( Site 1069), Richmond, Virginia
  - West Virginia University ( Site 1081), Morgantown, West Virginia
  - Aurora St Luke's Medical Center ( Site 1083), Milwaukee, Wisconsin
  - Froedtert Hospital & the Medical College of Wisconsin ( Site 1051), Milwaukee, Wisconsin
- Belgium (2):
  - Hôpital Erasme ( Site 1402), Anderlecht, Bruxelles-Capitale, Region de
  - UZ Leuven - Campus Gasthuisberg ( Site 1401), Leuven, Vlaams-Brabant
- Canada (4):
  - University Of Alberta ( Site 2101), Edmonton, Alberta
  - Hamilton General Hospital-Special Immunology Services Clinic ( Site 2110), Hamilton, Ontario
  - University Health Network ( Site 2109), Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie ( Site 2107), Sainte-Foy, Quebec
- France (12):
  - Hôpital Pasteur - CHU Nice ( Site 1311), Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire du Besancon ( Site 1324), Besançon, Doubs
  - Hopital de Rangueil du Toulouse ( Site 1322), Toulouse, Haute-Garonne
  - CHU Montpellier Hôpital Arnaud de VIlleneuve ( Site 1301), Montpellier, Herault
  - Hôpital Pontchaillou ( Site 1319), Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire de Grenoble ( Site 1303), Grenoble, Isere
  - CHU de Nantes - Hoptal Nord Laennec ( Site 1309), Nantes, Loire-Atlantique
  - CHU Angers ( Site 1313), Angers, Maine-et-Loire
  - CHRU de Nancy Hopitaux de Brabois ( Site 1308), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille ( Site 1306), Lille, Nord
  - CHU de Rouen ( Site 1323), Rouen, Seine-Maritime
  - Centre Hospitalier Universitaire de Bicetre ( Site 1304), Le Kremlin-Bicêtre, Val-de-Marne
- Germany (10):
  - Thoraxklinik-Heidelberg gGmbH ( Site 1509), Heidelberg, Baden-Wurttemberg
  - Krankenhaus Neuwittelsbach ( Site 1510), München, Bavaria
  - University Hospital Regensburg ( Site 1503), Regensburg, Bavaria
  - Kerckhoff-Klinik-Forschungs-GmbH ( Site 1514), Bad Nauheim, Hesse
  - Universitätsklinikum Gießen und Marburg GmbH ( Site 1512), Giessen, Hesse
  - Medizinische Hochschule Hannover ( Site 1505), Hanover, Lower Saxony
  - Uniklinik Köln ( Site 1511), Cologne, North Rhine-Westphalia
  - Universitaetsmedizin Johannes Gutenberg Universitaet Mainz ( Site 1515), Mainz, Rhineland-Palatinate
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden. ( Site 1501), Dresden, Saxony
  - DRK Kliniken Berlin Westend ( Site 1507), Berlin
- Israel (12):
  - Assuta Ashdod Medical Center ( Site 1710), Ashdod
  - Shamir Medical Center Assaf Harofeh ( Site 1713), Be’er Ya‘aqov
  - Rambam Health Corp. ( Site 1716), Haifa
  - Lady Davis Carmel Medical Center ( Site 1705), Haifa
  - Edith Wolfson Medical Center ( Site 1717), Holon
  - Shaare Zedek Medical Center ( Site 1715), Jerusalem
  - Hadassah Ein Kerem Medical Center ( Site 1711), Jerusalem
  - Meir Medical Center. ( Site 1707), Kfar Saba
  - Rabin Medical Center ( Site 1703), Petah Tikva
  - Kaplan Medical Center ( Site 1712), Rehovot
  - ZIV Medical Center ( Site 1704), Safed
  - Tel Aviv Sourasky Medical Center ( Site 1714), Tel Aviv
- Italy (7):
  - AOU di Bologna Policlinico S Orsola Malpighi ( Site 2409), Bologna, Emilia-Romagna
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) ( Site 2405), Trieste, Friuli Venezia Giulia
  - Fondazione IRCCS San Gerardo dei Tintori - ASST di Monza - A. O. San Gerardo ( Site 2406), Monza, Lombardy
  - Fondazione IRCCS-Policlinico San Matteo ( Site 2401), Pavia, Lombardy
  - Ospedale SS Annunziata ( Site 2408), Sassari, Sardinia
  - ASST Papa Giovanni XXIII ( Site 2410), Bergamo
  - Azienda Policlinico Umberto I ( Site 2402), Roma
- Unidad de Investigacion Clinica En Medicina SC ( Site 2505), Monterrey, Nuevo León, Mexico
- Poland (7):
  - Krakowski Szpital Specjalistyczny im Jana Pawla II ( Site 2801), Krakow, Lesser Poland Voivodeship
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego ( Site 2806), Lubin, Lublin Voivodeship
  - Europejskie Centrum Zdrowia Otwock Szpital im Fryderyka Chopina ( Site 2802), Otwock, Masovian Voivodeship
  - Państwowy Instytut Medyczny MSWiA ( Site 2805), Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku - Marii Sklodowskiej-Curie 24A ( Site 2803), Bialystok, Podlaskie Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie ( Site 2804), Szczecin, West Pomeranian Voivodeship
  - Wojewodzki Specjalistyczny Szpital im dr WI Bieganskiego w Lodzi ( Site 2807), Lodz, Łódź Voivodeship
- Spain (6):
  - Hospital Universitario Puerta de Hierro (Majadahonda) ( Site 1604), Majadahonda, Madrid
  - Hospital Costa del Sol ( Site 1613), Marbella, Malaga
  - Hospital Clinic de Barcelona ( Site 1602), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 1603), Madrid
  - Hospital Universitario Virgen Macarena ( Site 1612), Seville
  - Hospital Universitario de Toledo ( Site 1607), Toledo
- Sahlgrenska Universitetssjukhuset ( Site 3201), Gothenburg, Västra Götaland County, Sweden
- Imperial College Healthcare NHS Trust ( Site 1203), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26351&tenant=MT_MSD_9011